CLINICAL TRIAL: NCT04541316
Title: Neo-angiogenesis in 3D Dynamic Responsive Implant for Inguinal Hernia Repair ProFlor
Brief Title: Neo-angiogenesis in Inguinal Henia Implant ProFlor
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Giuseppe Amato, Consultant Professor, University of Cagliari
Other Study IDs: Neo-angiogenesis in ProFlor
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Inguinal Hernia
Keywords: Hernia implants; Biologic response; Neo-angiogenesis; Regenerative scaffolds
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue specimens excised from ProFlor prosthesis implanted in patients who underwent inguinal hernia repair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Short term post inguinal hernia repair with ProFlor: Determining presence and level of maturation of vascular structures in the inguinal hernia implant named ProFlor at 3-5 weeks post implantation
  Interventions: Device: ProFlor inguinal hernia device
- Mid term post inguinal hernia repair with ProFlor: Determining presence and level of maturation of vascular structures in the inguinal hernia implant named ProFlor at 3-4 months post implantation
  Interventions: Device: ProFlor inguinal hernia device
- Long term post inguinal hernia repair with ProFlor: Determining presence and level of maturation of vascular structures in the inguinal hernia implant named ProFlor at 6-8 months post implantation
  Interventions: Device: ProFlor inguinal hernia device

INTERVENTIONS:
Device: ProFlor inguinal hernia device — Inguinal hernia repair

SUMMARY:
The investigation is aimed at specifically demonstrating the ingrowth of newly formed vascular elements within ProFlor, a 3D dynamic responsive implant for inguinal hernia repair

DETAILED DESCRIPTION:
Biopsy specimen were excised at defined postoperative stages from patients who underwent hernia repair with the 3D prosthesis named ProFlor. Scope of the study was to determine the presence, quantity and quality of the vascular elements ingrowth within the implant fabric. Histology revealed the presence of multiple angiogenetic clusters that, starting from the early stage post-implantation, increased in number and degree of maturation. In the long term, the detected vascular components assumed the typical aspect of mature veins and arteries complete in all components. The development of fully developed vascular structures, ingrowing together with other components of the abdominal wall already described in literature, seems to finalize a regenerative response. This kind of behavior, being the expected result from a device intended for the cure of inguinal hernia and its degenerative source, seems to be coherent with the pathogenesis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent inguinal hernia repair with the 3D dynamic responsive device named ProFlor
* Patients undergoing recurrent inguinal hernia repair after primary repair with the 3D dynamic responsive device named ProFlor
* Patients undergoing surgical procedure in the groin area after inguinal hernia repair with the 3D dynamic responsive device named ProFlor

Exclusion Criteria:

* immunosoppressive therapy, > ASA 4 classification

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent inguinal hernia repair with the prosthetic device named ProFlor
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Ingrowth of Newly Formed Vascular Elements Within Hernia Implant ProFlor | 3-5 weeks post-implantation
  Post-operative assessment of neo-angiogenesis within hernia implant ProFlor at short term post-implantation
Ingrowth of Newly Formed Vascular Elements Within Hernia Implant ProFlor | 3-4 months post implantation
  Post-operative assessment of neo-angiogenesis within hernia implant ProFlor at midterm post-implantation
Ingrowth of Newly Formed Vascular Elements Within Hernia Implant ProFlor | 6-8 months post implantation
  Post-operative assessment of neo-angiogenesis within hernia implant ProFlor at midterm post-implantation

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Amato, Principal Investigator — University of Cagliari

IPD SHARING:
Plan to Share IPD: Yes
Tissue specimen and histological records upon request
Supporting Information: Study Protocol, SAP
Time Frame: from actual date until December 2022

REFERENCES:
- [Background] Amato G, Lo Monte AI, Cassata G, Damiano G, Romano G, Bussani R. A new prosthetic implant for inguinal hernia repair: its features in a porcine experimental model. Artif Organs. 2011 Aug;35(8):E181-90. doi: 10.1111/j.1525-1594.2011.01272.x. Epub 2011 Jul 13. PMID 21752035
- [Background] Amato G, Romano G, Agrusa A, Marasa S, Cocorullo G, Gulotta G, Goetze T, Puleio R. Biologic response of inguinal hernia prosthetics: a comparative study of conventional static meshes versus 3D dynamic implants. Artif Organs. 2015 Jan;39(1):E10-23. doi: 10.1111/aor.12416. PMID 25626584
- [Background] Amato G, Romano G, Puleio R, Agrusa A, Goetze T, Gulotta E, Gordini L, Erdas E, Calo P. Neomyogenesis in 3D Dynamic Responsive Prosthesis for Inguinal Hernia Repair. Artif Organs. 2018 Dec;42(12):1216-1223. doi: 10.1111/aor.13286. Epub 2018 Oct 14. PMID 30318605
- [Background] Amato G, Agrusa A, Puleio R, Calo P, Goetze T, Romano G. Neo-nervegenesis in 3D dynamic responsive implant for inguinal hernia repair. Qualitative study. Int J Surg. 2020 Apr;76:114-119. doi: 10.1016/j.ijsu.2020.02.046. Epub 2020 Mar 10. PMID 32169570
- See also: ProFlor inguinal hernia repair: features, procedural steps and clinical data — https://studio.youtube.com/channel/UCY7k5T6N3WtVqfTnitfTEfg/videos/upload?filter=%5B%5D&sort=%7B%22columnType%22%3A%22date%22%2C%22sortOrder%22%3A%22DESCENDING%22%7D